CLINICAL TRIAL: NCT03969186
Title: Use of A Telehealth Intervention to Decrease Readmissions in Cirrhosis: A Randomized Controlled Trial
Brief Title: Telehealth Intervention in Cirrhotics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 828183; chbgaidc (Other: University of Pennsylvania Institutional Review Board)
Record Dates: First submitted 2019-05-22; First posted 2019-05-31 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Cirrhosis, Liver; Liver Diseases
Keywords: Telehealth; Cirrhosis; Ascites; Hepatic encephalopathy; Readmissions; Preventable readmissions; Liver diseases; Variceal bleeding
MeSH Terms: conditions — Liver Cirrhosis; Liver Diseases; Fibrosis; Ascites; Hepatic Encephalopathy | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Daily telehealth follow-up (Experimental): The intervention arm will receive a simple telehealth intervention utilizing the Way to Health Platform engineered at the University of Pennsylvania. This platform will be used to send daily SMS messages to patients for 90 days following discharge and alert the research team to changes in patients' status. In addition, the patients in the intervention arm will receive a weekly phone call administered by members of the research team to assess their overall progress and well-being.
  Interventions: Behavioral: Intervention
- Standard of care follow-up (No Intervention): Standard of care

INTERVENTIONS:
Behavioral: Intervention — Telehealth intervention monitoring weight and medication adherence accompanied by a weekly phone call to monitor symptoms.
  Arms: Daily telehealth follow-up

SUMMARY:
This study is a randomized controlled trial comparing a simple telehealth intervention implemented after hospital discharge to standard of care, specifically looking at the number of hospital readmissions throughout the course of the study. All cirrhotic patients admitted to the Hepatology service at The Hospital of the University of Pennsylvania will be approached and consenting patients will be randomized to one of the two arms as outlined below. Patients will be followed for 90 days with daily texts and weekly phone calls. The rates of 30 and 90 day readmission as well as the days to readmission will be compared between the two study groups.

DETAILED DESCRIPTION:
Patients with cirrhosis and ascites comprise a large percentage of hospital admissions. As a large transplant center, the University of Pennsylvania sees an average of 54-65 cirrhotic patients admitted to the hepatology service every month. Many of these admissions are preventable and can be attributed to poor medication adherence and late detection of clinical deterioration. By introducing a telehealth intervention following hospital discharge, investigators seek to decrease the number of readmissions for these patients by encouraging and assisting with improved adherence and by regularly tracking the progression of symptoms.

This interventional study will serve a dual purpose of helping both the patient and their provider. Patients will obtain an extra line of communication to their providers that eases their ability to access resources and alert their providers to new symptoms. Similarly, by instituting a triaged system of communication with the patient, their health team is able to offer more individualized treatment while also providing more immediate attention at the first signs of clinical deterioration. This study will determine rates of 30 and 90-day readmissions in both cohorts as a way to examine the impact of a simple telehealth intervention compared to standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of cirrhosis of the liver
* Admitted to the Hospital of the University of Pennsylvania
* Ability to read and provide informed consent in English
* Ability to read and provide informed consent or surrogate present who can provide consent
* Possess a cell phone and willing to receive text messages.
* Has a surrogate who with a cell phone who is willing to receive and sent text messages for patient

Exclusion Criteria:

* Inability to provide informed consent in English
* Inability to provide informed consent or lack of surrogate who can provide consent
* Non-Cirrhotic
* Has received a liver transplant
* Discharged to hospice or has a disease process other than cirrhosis (i.e. severe heart disease or cancer) accounting for a high chance of mortality in the next 6 months.
* Advance symptoms of other disease process or too medically complex
* Actively using illicit substances or alcohol
* No access to cell phone with texting capability
* Not followed at the Hospital of the University of Pennsylvania

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2020-06-26 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
A change in readmission rates of cirrhotic patients | 90 Days
  Number of hospital readmissions during the 90 day intervention compared to control arm

SECONDARY OUTCOMES:
A difference in patient or caregiver satisfaction post-discharge. | 90 Days
  Self-reported patient satisfaction in surveys at 30 and 90 days looking at the research team's effectiveness, as well as provider communication. Satisfaction will be scored on a sliding scale and statistically analyzed to provide a quantifiable difference in satisfaction post-discharge for patients based on several aspects of their care.

CONTACTS AND LOCATIONS:
Overall Officials: Vandana Khungar, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- The Hospital of the University of Pennslyvania, Philadelphia, Pennsylvania, United States

DOCUMENTS (2):
  • Study Protocol (2018-09-26): https://cdn.clinicaltrials.gov/large-docs/86/NCT03969186/Prot_000.pdf
  • Informed Consent Form (2019-06-20): https://cdn.clinicaltrials.gov/large-docs/86/NCT03969186/ICF_002.pdf